CLINICAL TRIAL: NCT04485689
Title: The Effect of Capsaicin-induced Pain on Homeostatic Plasticity in Healthy Human Participants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aalborg University (Other)
Responsible Party: Principal Investigator, Priscilla G. Wittkopf, Principal Investigator, Aalborg University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: N-20190069/2
Record Dates: First submitted 2020-07-13; First posted 2020-07-24 (Actual); Last update posted 2020-08-31 (Actual); Status verified 2020-08

CONDITIONS: Healthy
MeSH Terms: interventions — Capsaicin

STUDY DESIGN:
Intervention Model Description: This is a within-between subjects comparisons study.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Capsaicin - alone (Experimental): 5x7 cm2 capsaicin patch
  Interventions: Drug: Capsaicin Topical - alone
- Placebo - alone (Placebo Comparator): 5x7 cm2 placebo patch alone
  Interventions: Drug: Placebo - alone
- Capsaicin - ice (Experimental): 5x7 cm2 capsaicin patch - plus ice
  Interventions: Drug: Capsaicin Topical - ice
- Placebo - ice (Placebo Comparator): 5x7 cm2 placebo patch - plus ice
  Interventions: Drug: Placebo - ice

INTERVENTIONS:
Drug: Capsaicin Topical - alone — 5x7 cm2 capsaicin patch applied on the dorsal area of the hand and left in place for 24 hours
  Arms: Capsaicin - alone
Drug: Placebo - alone — 5x7 cm2 patch applied on the dorsal area of the hand and left in place for 24 hours
  Arms: Placebo - alone
Drug: Capsaicin Topical - ice — 5x7 cm2 capsaicin patch applied on the dorsal area of the hand and left in place for 24 hours. Ice will be applied on top of the patch 1.5 hrs post patch application and left in place for 1 hr.
  Arms: Capsaicin - ice
Drug: Placebo - ice — 5x7 cm2 patch applied on the dorsal area of the hand and left in place for 24 hours. Ice will be applied on top of the patch 1.5 hrs post patch application and left in place for 1 hr.
  Arms: Placebo - ice

SUMMARY:
People suffering from chronic pain exhibit changes in the way the central nervous system processes pain. Some of the changes in the central nervous system are associated with how the brain adapts to the process of different stimuli. There are several physiological mechanisms that regulates how the brain adapts to changes and one of these mechanisms is called homeostatic plasticity (or equilibrium plasticity ). In healthy participants homeostatic plasticity mechanisms have been tested and considered normal, whereas in patients with chronic conditions, such as low back pain, this mechanism was shown to be dysfunctional. However, it is unknown when this difference in the pain system develops. It is possible that homeostatic mechanism becomes impaired during early stages of pain. This experiment will investigate the effect of capsaicin-induced pain on homeostatic plasticity in healthy participants.

DETAILED DESCRIPTION:
The aim of this study is to investigate the effect of capsaicin-induced pain on homeostatic plasticity.

A randomised crossover design will be used to evaluate the effect of capsaicin-induced pain on homeostatic plasticity using cathodal transcranial direct current stimulation (tDCS). Each participant will take part in four experimental sessions during which homeostatic plasticity and corticomotor excitability will be induced and measured in the left primary motor cortex. Participants will receive - in randomised order - capsaicin or placebo patch placed on the dorsal part of the right hand.

Each participant will attend four sessions, being two consecutive sessions separated by two weeks (i.e. wash-out period). During the experiment, participants will be seated comfortably with hands and arms at rest. First, the electromyography electrodes will be placed at the right first dorsal interosseous muscle to be used for assessing the corticomotor excitability by recordings of motor evoked potentials by transcranial magnetic stimulation (TMS) on the left primary motor cortex. Then, the cap for tDCS on the left primary motor cortex will be mounted. The optimal scalp position (hot spot) for TMS stimulation will be identified and marked with a pen on the cap for standardisation. A 5 x 7 cm capsaicin/placebo patch will be placed on participants' right hand. After 30 minutes of patch application, baseline measures of pain and motor-evoked potentials will be taken. Then, the homeostatic plasticity induction process will take place followed by motor-evoked potentials recordings every 15 minutes up to 45 minutes post protocol. Participants will be divided in 2 groups, one group will receive ice over the patch as to reduce pain intensity to minimum of 1 in a numeric rating scale; the other group will proceed without ice. Homeostatic plasticity will be induced and measured as previously described. The patch will be left in place for 24 hours, at which point participants will return to the laboratory and homeostatic plasticity will once again be induced and measured. After a wash-out period of two weeks, participants will go through an identical process but at this time with a different patch.

Homeostatic plasticity will be induced in the left primary motor cortex using tDCS applied for 7 minutes followed by an interval of 3 minutes and another block of 5 minutes of stimulation. A constant current of 2mA will be transmitted through the tDCS system, using two 25 cm2 electrodes placed into holes of a cap over the hot spot and right supraorbital area.

A sample size calculation was conducted using α of 0.05, β of 0.80 and effect size of 0.29 based on motor evoked potential (MEP) analysis of previous studies resulting in a target of 22 participants. To account for differences in designs 24 participants will be included, being 12 in each group.

Data distribution will be assessed using the Shapiro-Wilk test. A mixed analysis of variance (ANOVA) will be conducted on mean MEPs: within factors Intervention (Capsaicin and Placebo), Time (baseline, 0 min, 15 min, min, 30 min, 45 min), Time with pain (immediate, post pain relief post prolonged pain); and between factor (ice , no ice). A Greenhouse-Geisser correction will be used if Mauchly's test shows that sphericity cannot be assumed. Adjustments will be made for multiple post-hoc comparisons using the Bonferroni correction. Results will be interpreted according to the level of statistical significance p≤0.05.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, aged between 18-60 years, right-handed and can speak and understand English.

Exclusion Criteria:

* Lack of ability to cooperate
* Chili allergy
* History or present chronic pain or current acute pain
* Pregnancy
* Drug addiction defined as the use of cannabis, opioids or other drugs
* Present and previous neurological disorders such as epilepsy, Alzheimer's disease,
* dementia, stroke, migraine and other headache disorders, multiple sclerosis,
* Parkinson's disease, neuroinfections, brain tumors and head trauma.
* Present or previous musculoskeletal disorders such as tendonitis, degenerative disc disease, mechanical back syndrome, and ruptured/herniated disc.
* Present or previous mental illnesses such as depression, bipolar disorder, and schizophrenia.
* Current use of medications that may affect the trial (e.g. analgesics, anti- inflammatories, anti-depressives)
* Contraindications to TMS application (history of epilepsy, metal implants in head or jaw, etc.)
* Failure to pass the tDCS screening questionnaire
* Failure to pass the "TASS questionnaire"

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Conspiratorial excitability | [Time Frame: 0 minutes post homeostatic plasticity induction]
  Corticospinal excitability measured as motor evoked potentials amplitude induced by transcranial magnetic stimulation.
Conspiratorial excitability | [Time Frame: 15 minutes post homeostatic plasticity induction]
  Corticospinal excitability measured as motor evoked potentials amplitude induced by transcranial magnetic stimulation.
Conspiratorial excitability | [Time Frame: 30 minutes post homeostatic plasticity induction]
  Corticospinal excitability measured as motor evoked potentials amplitude induced by transcranial magnetic stimulation.
Conspiratorial excitability | [Time Frame: 45 minutes post homeostatic plasticity induction]
  Corticospinal excitability measured as motor evoked potentials amplitude induced by transcranial magnetic stimulation.

SECONDARY OUTCOMES:
Pain intensity | Every 10 minutes post capsaicin application
  Pain intensity measured using an 11-point numeric rating scale where 0= no pain and 10 = worst imaginable pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Aalborg University, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thapa T, Graven-Nielsen T, Chipchase LS, Schabrun SM. Disruption of cortical synaptic homeostasis in individuals with chronic low back pain. Clin Neurophysiol. 2018 May;129(5):1090-1096. doi: 10.1016/j.clinph.2018.01.060. Epub 2018 Feb 9. PMID 29472134
- [Background] Thapa T, Schabrun SM. Test-Retest Reliability of Homeostatic Plasticity in the Human Primary Motor Cortex. Neural Plast. 2018 Jun 10;2018:6207508. doi: 10.1155/2018/6207508. eCollection 2018. PMID 29983706
- [Background] Karabanov A, Ziemann U, Hamada M, George MS, Quartarone A, Classen J, Massimini M, Rothwell J, Siebner HR. Consensus Paper: Probing Homeostatic Plasticity of Human Cortex With Non-invasive Transcranial Brain Stimulation. Brain Stimul. 2015 May-Jun;8(3):442-54. doi: 10.1016/j.brs.2015.01.404. Epub 2015 Apr 1. PMID 26050599
- [Background] Fricke K, Seeber AA, Thirugnanasambandam N, Paulus W, Nitsche MA, Rothwell JC. Time course of the induction of homeostatic plasticity generated by repeated transcranial direct current stimulation of the human motor cortex. J Neurophysiol. 2011 Mar;105(3):1141-9. doi: 10.1152/jn.00608.2009. Epub 2010 Dec 22. PMID 21177994
- [Background] Rossini PM, Burke D, Chen R, Cohen LG, Daskalakis Z, Di Iorio R, Di Lazzaro V, Ferreri F, Fitzgerald PB, George MS, Hallett M, Lefaucheur JP, Langguth B, Matsumoto H, Miniussi C, Nitsche MA, Pascual-Leone A, Paulus W, Rossi S, Rothwell JC, Siebner HR, Ugawa Y, Walsh V, Ziemann U. Non-invasive electrical and magnetic stimulation of the brain, spinal cord, roots and peripheral nerves: Basic principles and procedures for routine clinical and research application. An updated report from an I.F.C.N. Committee. Clin Neurophysiol. 2015 Jun;126(6):1071-1107. doi: 10.1016/j.clinph.2015.02.001. Epub 2015 Feb 10. PMID 25797650